CLINICAL TRIAL: NCT06630143
Title: Effectiveness of Virtual Simulation Combined With Clinical Simulation in the Learning of Midwifery Students: A Randomized Clinical Trial
Brief Title: The Effectiveness of Combined Virtual and Clinical Simulation in Midwifery Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de los Andes, Chile (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Andrea López Navarrete, Professor, Universidad de los Andes, Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CEC2024016
Record Dates: First submitted 2024-09-24; First posted 2024-10-08 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Simulation Training; Midwifery Students Education; Clinical Competence; Education, Health; Virtual Simulation
Keywords: virtual simulation; clinical simulation; clinical judgment; randomized clinical trial; preeclampsia
MeSH Terms: conditions — Health Education; Pre-Eclampsia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessors (evaluators) will be blinded to the intervention groups (virtual simulation, clinical simulation, or combined simulation) to reduce potential bias in evaluating the study's outcomes. Assessors will evaluate participants; performance on theoretical knowledge and clinical judgment without knowing which intervention the participants received.
  Specifically, for the clinical judgment evaluation, the assessors will use the Lasater Clinical Judgment Rubric. The participants will be coded, and the assessors will only receive the coded evaluations to ensure they do not know the participants' group assignments. This blinding process will help ensure that the assessment of outcomes is objective and unbiased.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined Virtual and Clinical Simulation Arm (Experimental): Participants in this arm will receive a combination of virtual simulation using the vSim® platform and clinical simulation with a high-fidelity manikin. The virtual simulation focuses on the management of a preeclampsia case, which will be followed by a hands-on clinical simulation replicating the same scenario. This arm aims to assess whether combining both educational strategies enhances theoretical knowledge and clinical judgment more effectively than either method alone.
  Interventions: Other: Combined Virtual and Clinical Simulation
- Virtual Simulation Arm (Active Comparator): Participants in this arm will undergo a virtual simulation using the vSim® platform, which focuses on a preeclampsia case. This intervention will help participants develop clinical reasoning and decision-making skills in a virtual environment. The objective is to measure the effectiveness of virtual simulation alone on theoretical knowledge and clinical judgment.
  Interventions: Other: virtual simulation

INTERVENTIONS:
Other: Combined Virtual and Clinical Simulation — Participants will complete a preeclampsia case scenario through virtual simulation first and then engage in a clinical simulation involving the same case. This sequential intervention is designed to reinforce knowledge and skills.
  Arms: Combined Virtual and Clinical Simulation Arm
Other: virtual simulation — Participants will complete the preeclampsia case scenario using the vSim® platform, allowing them to engage in virtual clinical decision-making.
  Other Names: vSim
  Arms: Virtual Simulation Arm

SUMMARY:
Objective:

To evaluate the effectiveness of a combined virtual and clinical simulation strategy compared to virtual simulation alone and clinical simulation alone in the development of theoretical knowledge and clinical judgment among midwifery students, specifically in the management of preeclampsia.

Study Population:

75 undergraduate midwifery students in the second cycle of their studies at the Universidad de Los Andes, Chile.

Interventions:

Group 1: Virtual and Clinical Simulation combined (VSim® case on preeclampsia followed by hands-on clinical simulation with a manikin).

Group 2: Virtual Simulation only (VSim® case on preeclampsia).

Primary Outcomes:

Development of theoretical knowledge (measured by a test) on preeclampsia. Improvement in clinical judgment skills (assessed using the Lasater Clinical Judgment Rubric).

Secondary Outcomes:

Student satisfaction with the training. Perceived self-efficacy in managing preeclampsia. Usability of simulation platform

Duration:

The intervention lasts for 4 days. Pre- and post-tests will assess knowledge, clinical judgment, satisfaction, and self-efficacy.

Methodology:

A randomized controlled trial (RCT) with 35 participants divided equally into two groups. Each group will undergo either virtual simulation, or both. Data analysis will involve repeated measures ANOVA to assess the differences in learning outcomes between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment Status: Students in the second cycle of the midwifery program at the University of Los Andes.
* Educational Background: Participants must have completed the foundational courses in obstetrics and gynecology, as well as their initial clinical rotations.
* Consent: Participants must provide written informed consent to participate in the study.

Exclusion Criteria:

* Previous Clinical Experience: Students who have had prior clinical experience in high-risk obstetric units, or in preeclampsia management, will be excluded.
* Other Professional Backgrounds: Individuals with a degree or professional certification in obstetric or gynecological nursing (e.g., technicians with a title in obstetric nursing) will not be eligible.
* Exchange Students: Midwifery students participating in exchange programs will not be permitted to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Judgment in Managing Preeclampsia | Pre-intervention (before randomization) and post-intervention (Immediately after the assigned intervention).
  Clinical judgment will be evaluated using the Lasater Clinical Judgment Rubric (LCJR), a tool designed to assess the ability to observe, interpret, respond, and reflect in clinical situations. The rubric will be applied during a standardized clinical simulation scenario for preeclampsia management. The LCJR consists of 11 items, each rated on a scale from 1 to 4, for a total score ranging from 11 (minimum) to 44 (maximum). Higher scores indicate better clinical judgment and a more effective ability to manage clinical situations.
Theoretical Knowledge on Preeclampsia | Pre-intervention (before randomization) and post-intervention (Immediately after the assigned intervention).
  Theoretical knowledge will be assessed using a 10-item multiple-choice questionnaire specifically developed for this study, based on concepts from the American College of Obstetricians and Gynecologists (ACOG) and best practices for item construction. The test will be applied before and after the intervention to compare knowledge gains. The questionnaire will have a total score range of 0 (minimum) to 10 (maximum), with higher scores indicating better theoretical knowledge of preeclampsia.

SECONDARY OUTCOMES:
Satisfaction with the Learning Experience | Immediately after the assigned intervention
  The satisfaction of participants with the educational interventions will be measured using the Clinical Simulation Satisfaction Survey. This 15-item survey will use a 5-point Likert scale to gauge participants; satisfaction with the simulation activities. The scale ranges from 15 (minimum) to 75 (maximum). Higher scores indicate greater satisfaction with the educational interventions.
Perceived Self-Efficacy in Managing Preeclampsia | Pre-intervention (before randomization) and post-intervention (Immediately after the assigned intervention).
  Participants; perceived self-efficacy will be measured using the General Self-Efficacy Scale, validated for use in Chile. This scale contains 10 items rated on a 4-point Likert scale, assessing the participants' confidence in managing clinical situations like preeclampsia. The scale ranges from 10 (minimum) to 40 (maximum). Higher scores indicate greater perceived self-efficacy in managing clinical situations.
Usability of simulation platform | Immediately after the completion of the assigned intervention.
  The usability of the virtual and clinical simulation platforms will be assessed using the System Usability Scale (SUS), a widely used questionnaire that evaluates the ease of use, efficiency, and satisfaction with the simulation platforms. This outcome will provide insight into how user-friendly the simulation technologies are for midwifery students. The total SUS score ranges from 0 (minimum) to 100 (maximum), where higher scores indicate better usability. A SUS score above 68 is considered above average usability, while scores below that are considered below average.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de los Andes, Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No